CLINICAL TRIAL: NCT03162965
Title: Innovations in HIV Testing to Enhance Care for Young Women and Their Peers and Partners
Brief Title: Innovations in HIV Testing
Acronym: TI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Witwatersrand, South Africa (Other); University of California, San Francisco (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 15-1361b; 5R01HD083033 (NIH)
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants randomized to (1) Choice - they get to choose (1a) self-test vs (1b) HCT (HIV testing and counseling at clinic) or (2) they are randomized to HCT.
Oversight: Data Monitoring Committee: No | US Export: Yes

ARMS (2):
- Choice (Active Comparator): Oraquick HIV Self Test or Clinic Based HIV Counseling and Testing (HCT)
  Interventions: Other: Oraquick HIV Self Test; Other: Clinic Based HIV Counseling and Testing (HCT)
- HIV Counseling and Testing (Active Comparator): Clinic Based HIV Counseling and Testing (HCT)
  Interventions: Other: Clinic Based HIV Counseling and Testing (HCT)

INTERVENTIONS:
Other: Oraquick HIV Self Test — This is an oral swab in home HIV test.
  Arms: Choice
Other: Clinic Based HIV Counseling and Testing (HCT) — Receiving Counseling and Testing for HIV at the clinic.

SUMMARY:
The investigators propose to improve HIV prevention and care through expanding HIV testing options to include self-testing for young women, their peers and their sex partners, and by facilitating linkage to care.

DETAILED DESCRIPTION:
The investigators propose to improve HIV prevention and care through expanding HIV testing options to include self-testing for young women, their peers and their sex partners, and by facilitating linkage to care. In this study the investigators proposed two phases. The first phase, previously completed, is formative and involved two parts: 1) conducting formative qualitative research to understand perceptions of HIV testing and HIV self-testing in the study population and 2) conducting observed HIV self-testing to better understand any challenges with self-testing and the materials needed to make the process clear. The second phase of the study is a randomized controlled trial where the investigators will randomize approximately 400 young women to receive either 1) CHOICE of self-testing or clinic-based HIV Counseling and Testing (HCT) or 2) clinic based HCT. Once young women have been randomized, they will be asked to recruit up to 4 peers or male sex partners to test with the method of their randomization group.

ELIGIBILITY:
Eligibility Inclusion Criteria Index:

* Females ages 18-26
* Have had sex in the past 3 months and plan to have sex again in the next 3 months
* Planning on staying in the Agincourt Health and Demographic Surveillance System (AHDSS) area for the next nine months
* Able and willing to provide informed consent
* Willing to comply with study procedures
* Not known to be HIV positive (not reporting a previous positive test)

Eligibility Inclusion Criteria Peer/Partner:

* Females and Males ages 18 and older
* Able and willing to provide informed consent
* Willing to comply with study procedures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Enrolled participants need to self-identify as female. Peers and partners can be male and female.
Enrollment: 898 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Proportion of index reporting testing uptake | 3 months post randomization
  Compare between the two study arms the proportion of testing uptake at 3 months post-randomization. Testing uptake is defined for HCT as self-report of going to the clinic and testing; and for self-test as self-report of using a self-test kit.

SECONDARY OUTCOMES:
Proportion of peer/partner referrals by the index | 12 months post randomization
  Compare between the two studies arms the number of self test kits and HCT cards distributed by the index.
Proportion of peer/partners reporting testing uptake | 12 months post randomization
  Compare between the two study arms the proportion of testing uptake by peers/partners. Testing uptake is defined for HCT as self-report of going to the clinic and testing; and for self-test as self-report of using a self-test kit.
Proportion of index and peer/partners who obtain a confirmatory test, start Antiretroviral Treatment (ART) if HIV+, and obtain their Cluster of Differentiation 4 (CD4) count if HIV+ | 12 months post randomization
  Among participants who test positive (young women, peers and sex partners), the investigators will examine uptake of linkage to care.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Pettifor, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Medical Research Council/Wits University Rural Public Health and Health Transitions Research Unit, Acornhoek, Mpumalanga, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pettifor A, Lippman SA, Kimaru L, Haber N, Mayakayaka Z, Selin A, Twine R, Gilmore H, Westreich D, Mdaka B, Wagner R, Gomez-Olive X, Tollman S, Kahn K. HIV self-testing among young women in rural South Africa: A randomized controlled trial comparing clinic-based HIV testing to the choice of either clinic testing or HIV self-testing with secondary distribution to peers and partners. EClinicalMedicine. 2020 Apr 18;21:100327. doi: 10.1016/j.eclinm.2020.100327. eCollection 2020 Apr. PMID 32322811
- [Derived] Ritchwood TD, Selin A, Pettifor A, Lippman SA, Gilmore H, Kimaru L, Hove J, Wagner R, Twine R, Kahn K. HIV self-testing: South African young adults' recommendations for ease of use, test kit contents, accessibility, and supportive resources. BMC Public Health. 2019 Jan 29;19(1):123. doi: 10.1186/s12889-019-6402-4. PMID 30696422